CLINICAL TRIAL: NCT01718743
Title: Phase II Study of the Combination of MLN 9708 With Lenalidomide as Maintenance Therapy Post Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Ixazomib Citrate and Lenalidomide After Stem Cell Transplant in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0277; NCI-2012-02873 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0277 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate, lenalidomide) (Experimental): Beginning 60-180 days post-transplant, patients receive ixazomib citrate PO on days 1, 8, and 15 and lenalidomide PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib Citrate; Drug: Lenalidomide; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ixazomib citrate and lenalidomide after stem cell transplant work in treating patients with newly diagnosed multiple myeloma. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Giving ixazomib citrate together with lenalidomide may be effective in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish safety and efficacy of oral ixazomib citrate (MLN 9708) and lenalidomide in the maintenance setting post autologous stem cell transplant (ASCT) in myeloma patients.

SECONDARY OBJECTIVES:

I. Incidence of secondary primary malignancy.

II. Evaluate the best response rate (stringent complete response [sCR]/near complete response [nCR]/very good partial response [VGPR]/partial response [PR]).

III. Evaluate time to progression.

IV. Evaluate time to next therapy.

V. Evaluate the tolerability and toxicity.

VI. Evaluate M. D. Anderson Symptom Inventory (MDASI)-myeloma symptom evaluation.

OUTLINE:

Beginning 60-180 days post-transplant, patients receive ixazomib citrate orally (PO) on days 1, 8, and 15 and lenalidomide PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have undergone autologous stem cell transplantation, with melphalan as a preparative regimen, within 12 months of initiation of induction therapy for newly diagnosed myeloma
* Time to initiation of maintenance therapy; patients may start maintenance therapy as early as 60 days post-transplant and up to 180 days post-transplant; as long as they meet the following criteria:
* Platelet count >= 100,000/mm^3; platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Neutrophil count >= 1000/mm^3; (no growth factors within 5 days prior to first dose of the study drug)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine < 2.5 mg/dL
* Recovered (i.e., =< grade 1 toxicity) from the reversible effects of autologous stem cell transplant
* Patients whose primary therapy was changed due to suboptimal response of toxicity will be eligible, however no more than 2 regimens will be allowed prior to ASCT
* Patients must have an Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female patients who: are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR if they are childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent, during study treatment and for 90 days after the last dose of study treatment, AND

  * Must also adhere to guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following: agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study treatment, OR

  * Must also adhere to guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Major surgery within 14 days before the first dose of study drug
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708
* Known active central nervous system involvement
* Systemic treatment, within 14 days before study enrollment, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Female subject who are lactating or have a positive serum pregnancy test during the screening period
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation or completion of treatment according to this protocol
* Corrected QT interval using Bazett's formula (QTcB) > 470 milliseconds (msec) on a 12-lead electrocardiogram (ECG) obtained during the screening period; if a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG
* Ongoing or active systemic infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations
* Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krina Patel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 participants were enrolled in the study between December 3, 2012 and May 13, 2015
Pre-assignment Details: Participants with the following conditions were excluded from the study: grade 2 or higher peripheral neuropathy; major surgery or radiotherapy within 14 days of starting on the study; central nervous system involvement; treatment with modulators of CYP1A2 and CYP3A enzyme activity; and cardiovascular complications or ongoing systemic infections.
Groups:
- Treatment (Ixazomib Citrate, Lenalidomide): Beginning 60-180 days post-transplant, participants receive ixazomib citrate PO on days 1, 8, and 15 and lenalidomide PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Ixazomib Citrate: Given PO
  Lenalidomide: Given PO
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Started | 64
Completed | 19
Not Completed | 45
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 14
Not completed — Progressive Disease | 22
Not completed — Toxicity | 1
Not completed — Malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
Age, Customized [Number; unit: participants]
  Between 18-59 | 23
  >= 60 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Monitored using the method of Thall et al. Estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.
Time Frame: Time from autologous stem cell transplant (ASCT) to time of clinical progression or death or the time of last contact, assessed up to 30 days after completion of study treatment
Population: The upper bound of the 95% CI has not been reached.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
Months | 73.3 [59.9 to NA] — The upper bound of the 95% CI has not been reached.

2. Secondary Outcome: Best Response Rate (Stringent Complete Response [sCR]/Near Complete Response [nCR]/Very Good Partial Response [VGPR]/Partial Response [PR])
Description: Estimated along with 95% confidence intervals.
Time Frame: through out study treatment and up to 30 days after completion of study treatment, up to 119 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
percentage of participants | 98.4 [91.5 to 100]

3. Secondary Outcome: Treatment-related Unmanageable Toxicities, Including Grade 3 Non-hematologic Effects, or Grade 4 Hematologic Effects
Description: Toxicity data will be summarized by frequency tables.
Time Frame: throughout study treatment and up to 30 days after completion of study treatment, up to 119 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
Participants
  Serious AE-Lung Infections | 12
  Serious AE-Treatment-related secondary malignancy | 9
  Serious AE-Respiratory Disorders including respiratory failures | 8
  Serious AE-other infections | 5

4. Secondary Outcome: Number of Participants Incidence of New Primary Malignancy
Description: Count of participants
Time Frame: through out study treatment and up to 30 days after completion of study treatment, up to 119 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
Participants | 9

5. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method. Cox proportional hazards model will be used to include multiple covariates. Log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be used to include multiple covariates in the time-to-event analysis.
Time Frame: through out study treatment and up to 30 days after completion of study treatment, up to 119 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 64
months | NA [NA to NA] — The median OS time is the time point (from transplant) at which the probability of survival is 50%. If you look at the KM curve below for OS, the curve is going down overtime but has not reached the horizontal line for probability=0.5. The median OS time has not been reached. The 95% CI is not estimable.

6. Secondary Outcome: M. D. Anderson Symptom Inventory (MDASI)-Myeloma Symptom Evaluation
Description: Analyzed with descriptive analysis. The MDASI-MM scores measure the how severe the symptoms are, so higher scores are considered to be worse patient outcomes. Five subscales are derived from the 26 questions of the MDASI-MM questionnaire:
  1. mean core (13 MDASI core symptom items), ranges from 0 to 130.
  2. mean severity (13 MDASI core plus 7 MM-specific items), ranges from 0 to 200.
  3. mean interference (6 interference items), ranges from 0 to 60.
  4. mean WAW (interference with work, general activity, and walking), ranges from 0 to 30.
  5. mean REM (interference with relations with people, enjoyment of life, and mood), ranges from 0 to 30.
  has context menu
Time Frame: through out study treatment and up to 30 days after completion of study treatment, up to 119 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
Number analyzed (Participants) | 59
scores on a scale
  Core Score at Cycle 1 | 1.13 (1.35)
  Severity Score at Cycle 1 | 1.01 (1.27)
  Interference Score at Cycle 1 | 0.97 (1.52)
  WAW Score at Cycle 1 | 1.12 (1.67)
  REM Score at Cycle 1 | 0.81 (1.54)

ADVERSE EVENTS:
Time Frame: through out study treatment and up to 30 days after completion of study treatment, up to 119 months
Arm/Group | Treatment (Ixazomib Citrate, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 33/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ixazomib Citrate, Lenalidomide) (N=64)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 12
Respiratory, thoracic, and mediastinal disorders, including respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8
Infections and infestations (Infections and infestations) | 5
Treatment-related secondary malignancy (General disorders) | 9
Sepsis (General disorders) | 3
Neoplasms benign, malignant, and unspecified (inclcysts and ployps) (Blood and lymphatic system disorders) | 3
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Acute kidney inury (Renal and urinary disorders) | 1
Dehydration (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Fever (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
Nervous system disorders (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Syncope (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Lenalidomide) (N=64)
Abdomial pain (General disorders) | 5 (6)
Agitation (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (General disorders) | 35 (135)
Alkaline phosphatase increased (General disorders) | 21 (56)
Allergic reaction (General disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 27 (126)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (General disorders) | 2 (2)
Anxiety (Nervous system disorders) | 2 (3)
Arthralgia (General disorders) | 7 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Aspartate aminotransferase increased (General disorders) | 38 (146)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back Pain (General disorders) | 22 (41)
Bladder infection (Infections and infestations) | 1 (1)
Bloating (General disorders) | 4 (5)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 20 (22)
Blood bilirubin increased (General disorders) | 20 (228)
Blurred vision (Nervous system disorders) | 32 (114)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Breast pain (General disorders) | 1 (1)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 4 (5)
Cataract (General disorders) | 1 (1)
Chest pain (General disorders) | 3 (5)
Chills (General disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (3)
Conjunctivitis (Infections and infestations) | 2 (2)
Constipation (Gastrointestinal disorders) | 44 (258)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (40)
Creatinine increased (General disorders) | 29 (172)
Dehydration (General disorders) | 2 (3)
Depression (Nervous system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 53 (635)
Dizziness (Nervous system disorders) | 33 (168)
Dry eye (General disorders) | 31 (86)
Dry mouth (General disorders) | 12 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (14)
Dysgeusia (General disorders) | 3 (3)
Dyspepsia (General disorders) | 2 (3)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 36 (131)
Edema face (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (Skin and subcutaneous tissue disorders) | 37 (104)
Edema trunk (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders (General disorders) | 5 (6)
Eyelid function disorder (Nervous system disorders) | 1 (1)
Fall (General disorders) | 8 (10)
Fatigue (General disorders) | 60 (442)
Fever (General disorders) | 37 (103)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 8 (12)
Flushing (Vascular disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (5)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (9)
General disorders and administration site conditions (General disorders) | 2 (3)
Hallucinations (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (20)
Hearing impaired (Nervous system disorders) | 3 (4)
Hematuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (General disorders) | 16 (39)
Hyperglycemia (General disorders) | 43 (352)
Hyperkalemia (General disorders) | 13 (26)
Hypermagnesemia (General disorders) | 2 (2)
Hypernatremia (General disorders) | 5 (6)
Hypertension (General disorders) | 3 (3)
Hyperuricemia (General disorders) | 12 (24)
Hypoalbuminemia (General disorders) | 32 (85)
Hypocalcemia (General disorders) | 31 (130)
Hypoglycemia (General disorders) | 24 (79)
Hypokalemia (General disorders) | 28 (103)
Hypomagnesemia (General disorders) | 38 (165)
Hyponatremia (General disorders) | 5 (5)
Hypophosphatemia (General disorders) | 5 (7)
Hypotension (Vascular disorders) | 1 (2)
Infections and infestation (General disorders) | 29 (41)
Injury, poisoning and procedural complications (General disorders) | 1 (1)
INR increased (General disorders) | 1 (1)
Insomnia (Nervous system disorders) | 10 (13)
Investigations (General disorders) | 28 (51)
Lethargy (General disorders) | 1 (1)
Leukemia secondary to oncology chemotherapy (Blood and lymphatic system disorders) | 1 (1)
Lip Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 21 (30)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 22 (78)
Mania (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 31 (65)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 25 (182)
Mucositis oral (Skin and subcutaneous tissue disorders) | 23 (81)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 16 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 49 (209)
Nail infection (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 52 (474)
Neck pain (Nervous system disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (General disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 57 (814)
Non-cardiac chest pain (Nervous system disorders) | 1 (1)
Optic nerve disorder (Nervous system disorders) | 1 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Otitis media (Infections and infestations) | 2 (2)
Pain (Nervous system disorders) | 27 (51)
Pain in extremity (Nervous system disorders) | 7 (9)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 11 (17)
Peripheral sensory neuropathy (Nervous system disorders) | 54 (221)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Phlebitis infective (Vascular disorders) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 52 (284)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Prostate infection (Infections and infestations) | 1 (2)
Prostatic obstruction (General disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 10 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (32)
Psychiatric disorders (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (40)
Renal and urinary disorders (Renal and urinary disorders) | 7 (9)
Renal calculi (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders (General disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Scleral disorder (General disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Sinus disorder (Vascular disorders) | 1 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 16 (27)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 19 (24)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Spasticity (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Superficial thrombophlebitis (Blood and lymphatic system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 4 (4)
Tinnitus (Nervous system disorders) | 6 (9)
Tooth development disorder (General disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Infections and infestations) | 4 (4)
Tremor (Nervous system disorders) | 3 (3)
Upper respiraotry infection (Infections and infestations) | 41 (102)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 14 (23)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (2)
Vascular access complication (Vascular disorders) | 1 (1)
Voice alteration (General disorders) | 1 (1)
Vomiting (Nervous system disorders) | 41 (122)
Watering eyes (General disorders) | 26 (76)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WBC decreased (Blood and lymphatic system disorders) | 56 (748)
Wound complication (Skin and subcutaneous tissue disorders) | 1 (2)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT01718743/Prot_SAP_000.pdf